CLINICAL TRIAL: NCT01076439
Title: A Pilot Study Evaluating the Onset of Action of Fluticasone Furoate Nasal Spray and Olopatadine Nasal Spray Compared to Placebo Nasal Spray in Reducing Nasal Allergic Symptoms Following Ragweed Exposure in the Allergen BioCube (ABC)
Brief Title: An Allergen BioCube (ABC) Study Evaluating the Onset of Action of Fluticasone Furoate Nasal Spray and Olopatadine Nasal Spray Compared to Placebo
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10-270-0006
Record Dates: First submitted 2010-02-24; First posted 2010-02-26 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Olopatadine Nasal Spray (Patanase) (Active Comparator)
  Interventions: Drug: Olopatadine Nasal Spray
- Fluticasone Furoate Nasal Spray (Veramyst) (Active Comparator)
  Interventions: Drug: Fluticasone Furoate Nasal Spray
- Saline Nasal Spray (Placebo) (Placebo Comparator)
  Interventions: Drug: Saline Nasal Spray

INTERVENTIONS:
Drug: Fluticasone Furoate Nasal Spray — Fluticasone Furoate Nasal Spray: 110mcg QD
  Arms: Fluticasone Furoate Nasal Spray (Veramyst)
Drug: Olopatadine Nasal Spray — Olopatadine Nasal Spray: 2660mcg BID
  Arms: Olopatadine Nasal Spray (Patanase)
Drug: Saline Nasal Spray — Placebo
  Arms: Saline Nasal Spray (Placebo)

SUMMARY:
The purpose of this study is to evaluate the onset of action of fluticasone furoate nasal spray compared to olopatadine nasal spray and placebo nasal spray in reducing nasal allergic signs and symptoms following ragweed exposure in the Allergen BioCube (ABC) after single dose administration and six consecutive days of treatment.

ELIGIBILITY:
Inclusion Criteria:

* provide written informed consent and signed HIPAA form;
* be able and willing to follow all instructions and attend the study visits;
* if female and of childbearing potential, be not pregnant, nursing or planning a pregnancy, be willing to submit a pregnancy test at visit 1 and at exit visit, and to use adequate method of birth control
* have a positive history of seasonal allergic rhinitis to ragweed;
* have a positive skin test reaction to ragweed of within the past 24 months;
* manifest sufficient allergic rhinitis symptoms during ragweed exposure in the ABC

Exclusion Criteria:

* manifest symptoms of clinically active allergic rhinitis at the start of Visit 1 or Visit 2;
* known intolerance or allergy to antihistamines or corticosteroids;
* have a compromised lung function at Visit 1;
* have significant nasal anatomical deformities or any condition that does not allow subject to breathe through the nose (includes, but is not limited to: septal deviation, septal perforations, nasal polyps, rhinitis medicamentosa)
* have had any nasal surgical intervention in the past;
* have planned surgery (nasal, ocular or systemic) during the trial period or within 30 days thereafter;
* use disallowed medications (topical, topical ophthalmic, systemic and/or injectable treatments and all anti-allergy therapies including prescription, over the counter or homeopathy, and over the counter sleeping aids) during the study or appropriate pre-study washout period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Nasal Signs and Symptoms (TNSS) | Evaluated by the subject pre-ABC exposure, every 15 minutes during all ragweed exposures in the ABC, and post-ABC exposure
  TNSS (0-12 unit scale) is defined as the sum of the four nasal symptom scores recorded for nasal itching, sneezing, rhinorrhea and nasal congestion.

SECONDARY OUTCOMES:
Peak Expiratory Flow Rate (PEFR) | Measured pre-ABC exposure, every 30 minutes during all ragweed exposures in the ABC, and post-ABC exposure
Peak Nasal Inspiratory Flow (PNIF) | Measured pre-ABC exposure, every 30 minutes during all ragweed exposures in the ABC, and post-ABC exposure
Headaches | Evaluated by the subject pre-ABC exposure, every 30 minutes during all ragweed exposures in the ABC, and post-ABC exposure

CONTACTS AND LOCATIONS:
Overall Officials: H. J. Crampton, MD, Principal Investigator — ORA, Inc.